CLINICAL TRIAL: NCT03952247
Title: Prospective, Randomized Study in Ventilated Critically Ill Patients Receiving Percutaneous Tracheotomy. A Comparison of Periinterventional Visualization of Conventional Bronchoscopy and Single Use Bronchoscopy (TraSUB™)
Brief Title: "TRAcheostomy With Single Use Bronchoscopes vs. Conventional Bronchoscopes"
Acronym: TraSUB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TraSUB
Record Dates: First submitted 2019-04-28; First posted 2019-05-16 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Insufficiency
Keywords: tracheotomy; bronchoscopy; critical care
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Use Bronchoscopy (Experimental): optical guidance of percutaneous tracheotomy is done by single use bronchoscopy
  Interventions: Device: Single Use Bronchoscopy for PDT
- Conventional Multi Use Bronchoscopy (Active Comparator): optical guidance of percutaneous tracheotomy is done by conventional multi use bronchoscopy
  Interventions: Device: Conventional Multi Use Bronchoscopy for PDT

INTERVENTIONS:
Device: Single Use Bronchoscopy for PDT — optical guidance of percutaneous tracheotomy is done by single use bronchoscopy
  Arms: Single Use Bronchoscopy
Device: Conventional Multi Use Bronchoscopy for PDT — optical guidance of percutaneous tracheotomy is done by conventional multi use bronchoscopy
  Arms: Conventional Multi Use Bronchoscopy

SUMMARY:
Optical guidance for percutaneous tracheostomy in intensive care is usually performed by conventional multi use bronchoscopy. Recently a single use bronchoscope has been introduced that allows for endotracheal visualization.

For feasibility evaluation, 23 patients in intensive care receive percutaneous tracheostomy with optical guidance by the Ambu® aScopeTM 4 bronchoscope and 23 patients in intensive care receive percutaneous tracheostomy with a conventional bronchoscope (Olympus BF Type P60). The primary end point is the visualization through the single use bronchoscope of endotracheal landmark structures for tracheostomy and visualization of the needle insertion (according to score, see detailed description).

DETAILED DESCRIPTION:
Background Long-term ventilated critically ill patients often receive a tracheostomy to facilitate weaning from the ventilator and for prevention of secondary complications by the endotracheal tube. Besides surgical tracheostomy in which a muco-cutaneous fistula is prepared between trachea and outer skin, percutaneous tracheostomy (PDT) has been introduced, in which a cannula is being inserted into the trachea. After introduction of a guidewire, the trachea is then dilated. This intervention should be led by optical guidance, i. e. to verify the correct point of tracheal cannulation between the 2nd and 3rd tracheal cartilage and to minimize the risk for accidental injury to the membranous part of the trachea. Usually, optical guidance is performed by conventional multi use bronchoscopy. During bronchoscopy in ventilated patients, a drop in minute ventilation or an increase of carbon dioxide partial pressure with a consecutive respiratory acidosis may occur. Recently, a single use bronchoscope has been introduced that permits a continuous visualisation of the trachea on a monitor connected to the camera (Ambu® aScopeTM 4, Ambu, Ballerup, Denmark) . In this study, it is being evaluated whether the optical guidance during PDT can be performed by the Ambu® aScope 4. The advantage of a single use bronchoscope for percutaneous dilatative tracheostomy in comparison to a conventional reuseable bronchoscope is that there is no need for repair or decontamination after use.

Methods:

Design of Study/ No. of Patients:

Randomized, prospective study/ 46 patients With a sample size of 46 (randomized 1:1 in 2 groups of 23 each) a difference of 35% on a visualization score [6] may be seen with an α-error of 0,05 and a β-error of 1-0,8.

Procedures:

* screening for study inclusion according to inclusion and exclusion criteria.
* Percutaneous tracheostomy with Ciaglia Blue Rhino technique
* Visualization of PDT via a conventional multi use bronchoscope vs the aScopeTM 4 single use bronchoscope.

study inclusion: All patients being treated in the Dept. of Intensive Care Medicine receiving percutaneous tracheostomy due to long term ventilation are screened according to inclusion and exclusion criteria.

Details of study-procedures:

Bronchoscopy:

The bronchoscopy for percutaneous tracheostomy is done according to the standard operating procedure of the Dept. for Intensive Care Medicine. Furthermore, during this study the bronchoscopy is done by a physician with an experience of more than 200 bronchoscopies.

Percutaneous Tracheostomy:

The tracheostomy is performed according to the Ciaglia Blue Rhino method(Ciaglia Blue Rhino® G2, Cook Medical, Bloomington, IN, USA). After skin incision and an optional blunt dissection of the subcutaneous tissue, the trachea is cannulated between the 2nd and 3rd tracheal cartilage.

Visualization is provided by a conventional multi use bronchoscope or by a single use bronchoscope. Should visualization be insufficient by a single use bronchoscope backup is provided by a conventional multi use bronchoscope.

The tracheostomy is performed by an experienced fellow or attending physician. rating of visualization of tracheal structures and ventilation during percutaneous dilatational tracheostomy:

Rating (each item 1 to 4 points)

A) Identification of: thyroid cartilage, cricoid cartilage, 1st-3rd tracheal cartilage:

1 Reliable identification; 2 Only cricoid cartilage and tracheal cartilages; 3 Only tracheal cartilages; 4 No vision on tracheal structures

B) Visualization of tracheal circumference:

1 Complete; 2 circumference 1/3 to 2/3 of circumference; 3 Only small parts of trachea; 4 No vision on tracheal structures

C) Monitoring puncture: midline + level below 1st or 2nd tracheal cartilage:

1 Reliable identification; 2 Midline sure Level uncertain, but below the 1st tracheal cartilage; 3 Level of puncture uncertain; 4 No vision on tracheal structures

D) Monitoring dilatation Anterior wall and Pars membranacea (P.m.) visible:

1 Reliable identification; 2 P.m. only; 3 Only small parts of trachea visible, no control of P.m.; 4 No vision on tracheal structures

E) Quality of Ventilation Before puncture and worst ventilation during PDT, respectively:

1 Minute ventilation (MV) as before starting tracheotomy; 2 MV < 2 L/min or oxygen saturation (SO2) 80-90% (>2minutes); 3 MV < 0,5l /min or SO2 70 - 79% (> 2 minutes); 4 MV = 0 or SO2 < 70% (> 2 minutes)

F) Quality of the suction channel:

1 Uncomplicated suction of secretion; 2 suction only under flush; 3 suction only possible after multiple removing and flushing of the bronchoscope.; 4 suction not possible.

Consent: all patients or their legal surrogate give written informed consent.

Data protection: Data are anonymized.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving percutaneous tracheotomy in the Dept. of Intensive Care Medicine.
* Age ≥ 18 years
* Informed consent

Exclusion Criteria:

* Age < 18 years
* No consent
* Direct laryngoscopy according to Cormack-Lehane ≥ 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Visualisation | during tracheotomy
  visualisation through the single use bronchoscope of endotracheal landmark structures for tracheotomy and visualization of the needle insertion (according to score) Scale Name: Rating A) Identification of: thyroid cartilage, cricoid cartilage, 1st-3rd tracheal cartilage 1 Reliable identification; 2 Only cricoid cartilage and tracheal cartilages; 3 Only tracheal cartilages; 4 No vision on tracheal structures B) Visualization of tracheal circumference 1 Complete; 2 circumference 1/3 to 2/3 of circumference; 3 Only small parts of trachea; 4 No vision on tracheal structures C) Monitoring puncture: midline + level below 1st or 2nd tracheal cartilage
  1 Reliable identification; 2 Midline sure Level uncertain, but below the 1st tracheal cartilage; 3 Level of puncture uncertain; 4 No vision on tracheal structures D) Monitoring dilatation Anterior wall and Pars membranacea (P.m.) visible; 1 Reliable identification; 2 P.m. only; 3 Only small parts of trachea visible, no control of P.

SECONDARY OUTCOMES:
Minute ventilation | two time points: 1. during identification of landmark structures before puncture of trachea, 2. during puncture, dilatation and tracheotomy
  minute ventilation (according to score)
  Scale Name: Quality of Ventilation
  1 Minute ventilation (MV) as before starting tracheotomy; 2 MV < 2 L/min or oxygen saturation (SO2) 80-90% (>2minutes); 3 MV < 0,5l /min or SO2 70 - 79% (> 2 minutes); 4 MV = 0 or SO2 < 70% (> 2 minutes)
Peak airway pressure | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min after insertion of tracheal cannula
  changes in peak airway pressure of ventilator if volume controlled mode is used
  Measurement during following time Points:
  1. Measurements of Peak airway pressure before sterile drapes are applied; preintervention
  2. Measurement of Changes in Peak airway pressure before Skin incision and during identification of landmark structures
  3. Measure of Peak airway pressure after Insertion of the tracheal canula
pH | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min after insertion of tracheal cannula
  change in pH-values
  Measurement during following time Points:
  1. Measurements of pH values before sterile drapes are applied; preintervention
  2. Measurement of Changes in pH values before Skin incision and during identification of landmark structures
  3. Measurement of pH values after Insertion of the tracheal canula
paO2 | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min after insertion of tracheal cannula
  Change in paO2 values
  Measurement during following time Points:
  1. Measurements of paO2 values before sterile drapes are applied; preintervention
  2. Measurement of Changes in paO2 values before Skin incision and during identification of landmark structures
  3. Measurement of paO2 values after Insertion of the tracheal canula
paCO2 | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min after insertion of tracheal cannula
  Change in paCO2 values
  Measurement during following time Points:
  1. Measurements of paCO2 values before sterile drapes are applied; preintervention
  2. Measurement of Changes in paCO2 values before Skin incision and during identification of landmark structures
  3. Measurement of paCO2 values after Insertion of the tracheal canula
etCO2 | three time points: baseline value (before sterile drapes are applied), 0 min before skin incision, and 0 min after insertion of tracheal cannula
  Change in etCO2 values
  Measurement during following time Points:
  1. Measurements of etCO2 values before sterile drapes are applied; preintervention
  2. Measurement of Changes in etCO2 values before Skin incision and during identification of landmark structures
  3. Measurement of etCO2 values after Insertion of the tracheal canula
Duration of intervention | during tracheotomy (skin incision till insertion of tracheal cannula)
  Duration of Intervention
  Measurement of Duration of Intervention from Skin incision till Insertion of tracheal cannula (measured in minutes)
Poor visualisation | during tracheotomy
  Poor visualisation with single use bronchoscopy Poor identification thyroid cartilage, cricoid cartilage, 1st-3rd tracheal cartilage : Only identification of tracheal cartilages; No vision possible on tracheal structures Poor visualization of tracheal circumference: Only visualisation of small parts of trachea; No vision on tracheal structures
  Poor monitoring of puncture: midline + level below 1st or 2nd tracheal cartilage
  : Level of puncture uncertain; No vision on tracheal structures Poor Monitoring of Dilatation: Only small parts of trachea visible, no control of P.m.; No vision on tracheal structures
Poor control | during tracheotomy
  Poor control of the single use bronchoscope:
  Intubation of only one bronchial Segment not possible; Intubation of more than one bronchial Segment not possible.
adverse events | up to 1 week
  any adverse events that are likely associated with tracheostomy

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Grensemann, MD, Principal Investigator — Dept. of Intensive Care Medicine
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dreher M, Kluge S. [Airway devices in the intensive care unit]. Pneumologie. 2014 Jun;68(6):371-7. doi: 10.1055/s-0034-1365318. Epub 2014 Mar 25. German. PMID 24668495
- [Background] Ciaglia P, Firsching R, Syniec C. Elective percutaneous dilatational tracheostomy. A new simple bedside procedure; preliminary report. Chest. 1985 Jun;87(6):715-9. doi: 10.1378/chest.87.6.715. PMID 3996056
- [Background] Braune S, Kluge S. [Percutaneous dilatational tracheostomy]. Dtsch Med Wochenschr. 2011 Jun;136(23):1265-9. doi: 10.1055/s-0031-1280549. Epub 2011 May 31. No abstract available. German. PMID 21630175
- [Background] Vargas M, Sutherasan Y, Antonelli M, Brunetti I, Corcione A, Laffey JG, Putensen C, Servillo G, Pelosi P. Tracheostomy procedures in the intensive care unit: an international survey. Crit Care. 2015 Aug 13;19(1):291. doi: 10.1186/s13054-015-1013-7. PMID 26271742
- [Background] Grensemann J, Eichler L, Kahler S, Jarczak D, Simon M, Pinnschmidt HO, Kluge S. Bronchoscopy versus an endotracheal tube mounted camera for the peri-interventional visualization of percutaneous dilatational tracheostomy - a prospective, randomized trial (VivaPDT). Crit Care. 2017 Dec 29;21(1):330. doi: 10.1186/s13054-017-1901-0. PMID 29284503
- [Background] Baumann HJ, Kemei C, Kluge S. [Tracheostomy in the intensive care unit]. Pneumologie. 2010 Dec;64(12):769-76. doi: 10.1055/s-0030-1255743. Epub 2010 Sep 20. German. PMID 20857374
- [Background] Byhahn C, Wilke HJ, Halbig S, Lischke V, Westphal K. Percutaneous tracheostomy: ciaglia blue rhino versus the basic ciaglia technique of percutaneous dilational tracheostomy. Anesth Analg. 2000 Oct;91(4):882-6. doi: 10.1097/00000539-200010000-00021. PMID 11004042
- [Background] Linstedt U, Zenz M, Krull K, Hager D, Prengel AW. Laryngeal mask airway or endotracheal tube for percutaneous dilatational tracheostomy: a comparison of visibility of intratracheal structures. Anesth Analg. 2010 Apr 1;110(4):1076-82. doi: 10.1213/ANE.0b013e3181d27fb4. PMID 20357150
- [Derived] Tariparast PA, Brockmann A, Hartwig R, Kluge S, Grensemann J. Percutaneous dilatational tracheostomy with single use bronchoscopes versus reusable bronchoscopes - a prospective randomized trial (TraSUB). BMC Anesthesiol. 2022 Apr 2;22(1):90. doi: 10.1186/s12871-022-01618-4. PMID 35366806